CLINICAL TRIAL: NCT02741024
Title: In Vivo Efficacy of Artesunate-amodiaquine and Artemether-lumefantrine for the Treatment of Uncomplicated Falciparum Malaria: an Open-randomised, Non-inferiority Clinical Trial in South Kivu, DR Congo
Brief Title: Efficacy of Artesunate-amodiaquine and Artemether-lumefantrine for Uncomplicated Malaria in South Kivu, DR Congo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Principal Investigator, Marit de Wit, Health Advisor, Medecins Sans Frontieres, Netherlands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSansFrontieres
Record Dates: First submitted 2015-12-11; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amodiaquine-Artesunate (ASAQ) (Active Comparator): Treatment regimen consisted of Amodiaquine-Artesunate (ASAQ) fixed dose (FD) (Winthrop Sanofi Aventis), given as 1 tablet/day 3 days (5-8 kg 1 tab of 25mg artesunate/67.5 mg amodiaquine base, 9-17 kg 50 mg artesunate/135 mg amodiaquine base)
  Interventions: Drug: Amodiaquine-Artesunate (ASAQ)
- Artemether-Lumefantrine (AL) (Active Comparator): Treatment consisted of Artemether-Lumefantrine (AL) (Coartem, Novartis) given as six twice/daily doses over three days (5-14 kg 1tab of 20mg artemether/120mg lumefantrine BD, 15-24 kg 2tabs of 20mg artemether/120mg lumefantrine BD with fatty food).
  Interventions: Drug: Artemether-Lumefantrine (AL)

INTERVENTIONS:
Drug: Amodiaquine-Artesunate (ASAQ) — Treatment on site with Amodiaquine-Artesunate according to the manufacturer's dose and instruction and follow-up for a period of 42 days. Drugs will be given under direct supervision, either at the clinic or at home
  Other Names: coarsucam
  Arms: Amodiaquine-Artesunate (ASAQ)
Drug: Artemether-Lumefantrine (AL) — Treatment on site with Artemether-lumefantrine combination according to the manufacturer's dose and instruction and follow-up for a period of 42 days.
  Other Names: coartem
  Arms: Artemether-Lumefantrine (AL)

SUMMARY:
This will be an open-randomised non-inferiority study to test the hypothesis that the risk of recurrent parasitaemia after 42 days is not worse in the group receiving the Artesunate-Amodiaquine (ASAQ) regimen than in the group receiving the Artemether-Lumefantrine (Coartem®) regimen. Children with uncomplicated malaria meeting the inclusion criteria will be enrolled (after their parent/caretaker has given informed consent), treated on site with the drugs under evaluation and followed-up for a period of 42 days. Drugs will be given under direct supervision, either at the clinic or at home. Follow-up shall consist of a fixed schedule of clinical and laboratory examinations. Based on clinical and laboratory findings, children will be classified as therapeutic failures (early or late) or adequate responders.

The proportion of cases experiencing an in vivo therapeutic failure during the follow-up period will provide an estimate of the efficacy of the drug regimens. A Polymerase Chain Reaction (PCR) analysis will be carried out to differentiate true recrudescence due to treatment failure from episodes of re-infection. This proposal is compliant with the latest WHO recommendations for anti-malarial efficacy monitoring in high, medium or low transmission zones11.

DETAILED DESCRIPTION:
3.1 STUDY DESIGN Children with uncomplicated malaria meeting the inclusion criteria will be enrolled (after their parent/caretaker has given informed consent), treated on site with the drugs under evaluation and followed-up for a period of 42 days. Drugs will be given under direct supervision, either at the clinic or at home. Follow-up shall consist of a fixed schedule of clinical and laboratory examinations. Based on clinical and laboratory findings, children will be classified as therapeutic failures (early or late) or adequate responders.

The proportion of cases experiencing an in vivo therapeutic failure during the follow-up period will provide an estimate of the efficacy of the drug regimens. A Polymerase Chain Reaction (PCR) analysis will be carried out to differentiate true recrudescence due to treatment failure from episodes of re-infection. This proposal is compliant with the latest WHO recommendations for anti-malarial efficacy monitoring in high, medium or low transmission zones11.

3.2 STUDY SITES The study site will be the MSF catchment area of Baraka health centres, MSF-OCA Baraka, South Kivu, DRC.

3.3 STUDY POPULATION The study population is children aged between 6 and 59 months with uncomplicated P. falciparum malaria. This age group was selected because it is considered the most vulnerable and is less likely to clear infections spontaneously compared to older children and adults. In hyper-endemic areas, they are the most at risk of dying from malaria.

3.4 DEFINITIONS 3.4.1 DEFINITION OF PARENT/CARETAKER The parent/caretaker is defined as the household member who is aged ≥ 18 years who cares for the patient and can give accurate information on all demographic and health issues related to the patient and is present at the time of the survey.

3.5 INCLUSION AND EXCLUSION CRITERIA

A child will be eligible for study participation if s/he meets all of the following inclusion criteria:

* Age between 6 and 59 months
* Weight ≥ 5 Kg
* Slide-confirmed infection with Plasmodium falciparum only (no mixed infections)
* Asexual parasite density between 2000 and 200000/µl of blood
* Measured axillary temperature ≥ 37.5°C
* Ability to swallow oral medication
* High probability of respecting the follow-up visits (residence within 1 hour walking distance from the OPD, no upcoming travel plans, etc.)
* Informed consent from a parent or caretaker aged at least 18 years.

A child will be excluded from study participation if s/he meets any of the following exclusion criteria:

* General danger signs according to the WHO definition (Appendix 5.1.1)
* Signs of severe/complicated malaria according to the WHO definition (Appendix 5.1.2)
* Severe anaemia (haemoglobin < 5 g/dL)
* Known history of hypersensitivity to any of the study drugs
* Severe acute malnutrition (as defined by a weight-for-height below -3 Z-score and/or symmetrical oedemas involving at least the feet)
* Concomitant febrile illness due to causes other than malaria with the potential to confound study outcome (measles, acute lower tract respiratory infection, otitis media, tonsillitis, abscesses, severe diarrhoea with dehydration).
* Having received already a full course of the treatment (or one of the treatments) under study in the previous 28 days (as indicated by the parent/caretaker). Note that previous incomplete anti-malarial intake of treatments under study, or previous intake of anti-malarials not under study, are not exclusion criteria, but details of any such intake should be recorded carefully.
* History of hypersensitivity reactions or contra-indications to any medicines being tested.

3.6 SAMPLE SIZE Recent studies had determined the 42-day risk of recurrent parasitaemia due to recrudenscence (treatment failure) in children to range from 0.9-6% with Coartem® therapy14;17;21;22. Therefore on the basis of a conservative estimated risk of recurrent parasitaemia (due to recrudescence, PCR corrected) of 5%, we calculated that 120 patients per treatment arm would be needed to detect a difference in the risk of recurrent parasitaemia between treatment arms of no greater than 7% (one-sided type I error of 5%, 80% power)23.

Assuming re-infections, undetermined PCR results or loss to follow-up occur in 20% of samples, the total estimated sample size of this study will be 288 children aged 6-59 months (144 per arm).

3.7 SCHEDULE OF ASSESSMENTS Day 0 is the day of screening with clinical assessment, initial malaria blood smear, first haemoglobin measurement, pre-treatment capillary blood sample for PCR, enrolment and administration of first dose of drugs under study. On Day 1 and Day 2, treatment will continue and children will be re-assessed at the MSF clinic.

Children will return to the clinic on the following mandatory days: Day 3, 7, 14, 21, 28, 35 and 42. At each scheduled visit, a clinical examination and a blood smear will be performed. To encourage clinic attendance, small incentives will be offered such as soap, blankets and travel reimbursement. All children recruited to the study receive a long-lasting insecticide-treated bednet.

If children have to return to the clinic for unscheduled visits, at each time clinical and laboratory exams will be conducted as needed. In case of treatment failure at any day after day 7, a capillary blood sample for PCR will be collected.

3.8 STUDY END POINTS A study endpoint is the point at which a patient will no longer be followed-up within the context of the efficacy study. Valid study endpoints include treatment failure, completion of the follow-up period without treatment failure, loss to follow-up, withdrawal from study (voluntary and involuntary) and protocol violation11.

3.8.1 EARLY TREATMENT FAILURE (ETF)

* Development of danger signs or severe malaria on Day 1, Day 2 or Day 3 in presence of parasitaemia , or
* Parasitaemia on Day 2 higher than Day 0 count irrespective of axillary temperature, or
* Parasitaemia on Day 3 with axillary temperature ≥ 37.5°C, or
* Parasitaemia on Day 3 ≥ 25% of day 0 count irrespective of axillary temperature.

3.8.2 LATE CLINICAL FAILURE (LCF)

* Development of danger signs or severe malaria on any day from Day 4 to Day 42 in the presence of parasitaemia (without previously meeting any of the criteria of ETF), or
* Presence of parasitaemia and axillary temperature ≥ 37.5°C on any day from Day 4 to Day 42 (without previously meeting any of the criteria of ETF) 3.8.3 LATE PARASITOLOGICAL FAILURE (LPF)
* Presence of parasitaemia and axillary temperature < 37.5°C on any day from Day 7 to Day 42 (without previously meeting any of the criteria of ETF or LCF) 3.8.4 ADEQUATE CLINICAL AND PARASITOLOGICAL RESPONSE (ACPR)
* Absence of parasitaemia on Day 42 irrespective of axillary temperature (without previously meeting any of the criteria of ETF, LCF or LPF) 3.8.5 NON ANALYSABLE ENDPOINTS A patient's endpoint is not analysable if s/he meets any of the following criteria after his enrolment in the study. In non-inferiority studies, Intention-to-treat (ITT) analysis will often increase the risk of falsely claiming non-inferiority (type I error) so will not be carried out here24.

3.8.5.1 Protocol violation:

* Failure to complete the full study treatment regimen, other than due to vomiting,
* Erroneous enrolment of the patient (not all inclusion/exclusion criteria respected),
* Intake of any anti-malarials or antibiotics with anti-malarial activity (cotrimoxazole, tetracycline except for eye ointment, doxycycline, erythromycin, clindamycin, azithromycin) as administered by a third party or through self-medication,
* Misclassification of the patient's endpoint (due to a laboratory or clinical error) leading to the unjustified administration of the rescue treatment,
* LCF or LPF with missing or undetermined PCR result. 3.8.5.2 Withdrawal:
* Severe malaria occurring on Day 0 after enrolment,
* Detection of a (mixed or mono-) infection with a non-falciparum species,
* Vomiting any study dose more than once,
* Side effects of the study drug severe enough that they require discontinuation of treatment,
* Hospitalisation for a reason other than malaria, rendering normal follow-up visits impossible.
* Withdrawal of consent

3.8.6 SAFETY ENDPOINTS The occurrence of any adverse event will be documented. All patients will be asked routinely about previous symptoms and about symptoms that have emerged since the previous follow-up visit. When clinically indicated, patients will be evaluated and treated appropriately. All serious adverse events will be recorded on the case report form.

3.9 STUDY TREATMENTS 3.9.1 REGIMENS TESTED

* Artesunate-amodiaquine fixed dose combination, ASAQ FDC (artesunate-amodiaquine Winthrop® Sanofi Aventis) given as 1 tablet/day for 3 days:

  * Artesunate 25mg / amodiaquine 67.5mg: in children 5 to 8.9kg
  * Artesunate 50mg / amodiaquine 135mg: 1 tab/day in children 9 to 17.9kg
  * Artesunate 100mg / amodiaquine 270mg: 1 tab/day in children 18 to 34.9kg
* Artemether 20mg / lumefantrine 120mg co-formulated tablets (Coartem®, Novartis) given as six twice-daily doses over three days:

  * 1 tab/dose for children 5 to 14.9kg (total 6 tabs)
  * 2 tabs/dose for children 15 to 24.9kg (total 12 tabs)
  * 2 tabs/dose for weight 15-24.9kg (total 12 tabs)
  * 3 tabs/dose for weight 25-34.9 Kg (total 18 tabs) The second dose of Coartem® will be given 8 hours (h) after the first dose, given at enrolment. The following doses will be given 24h, 36h, 48h and 60h after the first dose. Patients will be given a glass of milk or fatty food, or encouraged to breastfeed before each dose is taken.

Drugs under study will come from the same batch. All study doses will be supervised. Patients will be directly observed following intake for 30 minutes. If vomiting occurs, a repeat dose will be administered. If the repeated dose is also vomited, the child will be withdrawn from the study, and rescue treatment will be initiated.

In order to administer the evening doses of Coartem®, a home visitor/village health worker will go to the patient's home 8h, 32h and 56h after the first dose. Thus recruitment to this study will only take place in the OPD before 12pm 3.9.2 CONCOMITANT TREATMENT Fever over 38°C can be treated with paracetamol or acetaminophen, one dose of 20 mg/kg of paracetamol, followed with 15 mg/kg at 4 to 6 hourly intervals for home treatment. Tepid sponging can be used to reduce fever before drug intake.

Adverse events requiring treatment can be treated according to local prac¬tice. If there is a clinical indication for any additional medication during the course of the study, including medication given to treat an adverse event related to the study medicine, the name of the medicine, the dosage and the date and time of administration must be recorded on the case report form. Additional prescriptions may be given on enrolment or during follow-up for conditions other than malaria, although antibiotics with anti-malarial activity (cotrimoxazole, tetracycline except for eye ointment, doxycycline, erythromycin, clindamycin, azithromycin) will not be prescribed unless no equally effective alternatives are available. Any such prescriptions will be noted carefully.

The use of herbal remedies during the study should be avoided, and partici¬pants should be encouraged to return to the study site for treatment if they feel unwell. If any herbal remedies are taken during the study, this should be captured on the case report form, under 'study medication administration'.

Haematinics (like ferrous sulphate and folic acid) will be prescribed to ameliorate anaemia according to WHO25 if necessary.

3.9.3 RESCUE TREATMENT

Rescue treatment for malaria shall be initiated immediately according to WHO guidelines25 for the following cases:

* Progression to severe malaria on Day 0 after enrolment
* Vomiting any study dose more than once
* Early treatment failure
* Late clinical failure
* Late parasitological failure
* Detection during follow-up of a non-P. falciparum (mixed or mono-) infection, irrespective of fever Rescue treatment shall consist of six-dose Coartem® for 3 days for the children that had received ASAQ as study-treatment or ASAQ for the children that had received Coartem® as study-treatment.
* In cases of severe malaria, rescue treatment will be intravenous artesunate at a dose of 2.4 mg/kg at 0, 12 and 24 hours, then once every 24 hrs until the patient can take oral therapy (This will be followed by 3-days full course of ACT) Non-falciparum species detected during follow up should be treated with Chloroquine for 3 days in the case of infection with P. vivax or P. ovale.

Once rescue treatment is initiated, normal study follow-up ends for the patient, as an endpoint has been reached. However, patients who receive rescue treatment will be asked to return to the study clinic at least once, so that the study team can verify whether the treatment has been effective.

3.10 STUDY PROCEDURE 3.10.1 SCREENING AND ENROLMENT (DAY 0) All children aged between 6 and 59 months presenting at the Baraka Health clinic with fever or a history of fever and positive RDT and with no danger signs (Appendix 5.1.1) will be sent to the study clinic for screening.

All patients entering the screening process will be assigned a consecutive screening number. The screening form (Appendix 5.2) will be used to record the general information and the clinical observations of each patient being screened. Each patient will be assessed again for danger signs and signs of severe malaria. Middle-upper arm circumference (MUAC) will then be used as a screening tool for malnutrition. An initial clinical assessment will be done including inclusion and exclusion criteria, previous treatment history (including ingestion of any anti-malarial drugs), clinical examination and weight-for-height on children with MUAC <125 mm.

Care will be taken to detect early signs of febrile diseases other than malaria, as their presence will necessitate exclusion from the study. These patients will not be enrolled but should be treated for both malaria (if they have parasitaemia) and the other infection, as appropriate.

If the patient meets the clinical inclusion criteria, s/he will be examined for blood inclusion criteria (P. Falciparum mono-infection, parasite density and haemoglobin levels). Thick and thin malaria smears will be taken on the same slide in duplicate and one smear will be stained. At the same time, a capillary blood sample will be taken on Fast Technology for Analysis (of nucleic acids) or FTA Cards for PCR analysis. The patient will wait for the thick smear result.

If all inclusion criteria are met, the patient will be invited to enrol in the study. The study purpose will be explained to the parent/caretaker who must be aged 18 years or above and a written informed consent will be requested (Appendix 5.4). All parents/caretakers will receive an information sheet containing the study purpose and study team contact details (Appendix 0).

If the parent/caretaker consents to include the child in the study, a unique patient identification number will be assigned to the child and a wrist band with the identification number will be given. Administrative data will be recorded (name of child and parent/caretaker, gender, age, address and directions) on a Case Record Form (Appendix 5.5). An appointment schedule will be clearly explained and a follow-up card marked with the unique patient identification number will be handed out.

Each unique patient identification number will be randomised to a treatment regimen before the study starts and this information will be contained in sealed envelopes. The first dose of the study drug will be dispensed at the health clinic (for children who cannot swallow, Coartem® tablets will be dissolved, and ASAQ tablets will be crushed in minimal amounts of water and dispensed by help of a syringe or dropper). Intake will be observed for 30 minutes. If the child vomits, a resting period of 15 minutes will be observed before attempting a repeat dose. Any concomitant prescriptions will be collected at the designated pharmacy and care will be taken to ensure that the instructions on home treatment are clear to the parent/caretaker.

Before being sent home, the patient's parent/caretaker will repeatedly be advised to bring him/her back the study clinic at any time if symptoms persist or worsen.

In order to administer the evening doses of Coartem®, a home visitor/village health worker will go to the patient's home 8h, 32h and 56h after the first dose. Thus recruitment to this study will only take place in the OPD before 12pm.

3.10.2 FOLLOW-UP (DAY 1 TO DAY42) On Days 1 and 2, study drug treatment is continued; the fourth (Day 1) and sixth (Day 2) Coartem® doses will be administered at home as described above by a home visitor. However all patients will return to the MSF clinic for a clinical assessment (including measurement of axillary temperature) and parasitological examination by malaria slide. All ASAQ and the 3rd and 5th Coartem® doses will be observed during these clinic visits.

On Days 3, 7, 14, 21, 28, 35 and 42, all patients will return to the MSF clinic for a clinical assessment (including axilliary temperature) and blood smear examination.

If treatment failure is observed (ETF, LCF or LPF) rescue treatment will be initiated. For LCF or LPF occurring after Day 7 (since if there is a re-infection it will not lead to clinical symptoms before day 7 so we can assume it's a recrudescence) a second blood sample will be collected on FTA cards for PCR analysis.

For unscheduled visits by patients, a clinical assessment will be performed, and a malaria slide (and blood sample for PCR in case of treatment failure) may be taken if there are signs and symptoms of possible malaria.

Before being sent home after each visit, the parent/caretaker will be advised to bring the patient back to the MSF clinic at any time in case of any illness. In case of emergency outside of working hours, parents/caretakers will be advised to bring their appointment card and to inform emergency staff of their child's inclusion in the study.

Instructions will be given to emergency staff to report all information concerning the event to the study coordinator the next morning.

Attempts to trace children who fail to return for scheduled visits will be made immediately by a home visitor to minimise loss to follow-up.

Patients who fail to return on days 1 and 2 and miss one dose of the treatment will be withdrawn from the study. After day 3, patients who fail to return on day 7 but are present on day 6 or 8 (likewise days 13/15, days 20/22, days 27/29, days 34/36 and days 41/43) may still be included in the analysis.

3.10.3 MEASUREMENT TECHNIQUES

* Weight will be measured to the nearest 100 g on a hanging scale (Salter) properly calibrated with only undergarments kept on the child.
* Height will be measured on a wooden height board, by asking the child to stand if s/he is > 85 cm, or by laying the child horizontally if s/he is < 85 cm.
* MUAC will be measured on the left arm, at the mid-point between the elbow and the shoulder and will be recorded to the nearest mm.
* Oedema will be assessed by 3 second thumb pressure on the dorsal surface of both feet.
* Axillary temperature will be measured with a calibrated digital thermometer graduated in Celsius, with a precision of 0.1°C. If the result is <36.0°C, the measurement will be repeated.

3.11 LABORATORY TECHNIQUES 3.11.1 MALARIA SLIDES

Thick and thin smears will be prepared on the same slide and stained in 10% Giemsa solution (pH 7.2) for 10-15 minutes. All smears must be read to 100 fields before they can be declared negative. Species will be confirmed on the thin smear. Quantification of P. falciparum asexual parasitaemia on the thick smear will be performed according to the WHO protocol26. Parasites will be counted against at least 200 white blood cells/leucocytes (WBC), and the parasite density (expressed in parasites per µL of blood) will be calculated assuming a normal level of 8000 WBC/µL:

Parasite density (/µL) = number of parasites counted x 8000 / number of WBC counted If 500 parasites are counted before reaching 200 WBC, the counting will be stopped at the end of that field and the parasitaemia will be calculated with the above formula. If less than 10 parasites are counted after 200 WBC, the counting will be extended to 500 white cells.

Presence or absence of P. falciparum gametocytes does not influence endpoint classification, but will be recorded carefully and systematically. If a smear contains gametocytes but not trophozoites (asexual parasites) it will be considered negative.

Two qualified microscopists will read all the slides independently, and parasite densities will be calculated by averaging the two counts. Blood smears with discordant results (differences between the two microscopists in species diagnosis, in parasite density of >50% or in the presence of parasites) will be re-examined by a third, independent microscopist and parasite density will be calculated by averaging the two closest counts.

All blood smears will be destroyed once data analysis is complete. 3.11.2 HAEMOGLOBIN MEASUREMENT The HemoCue B-Haemoglobin analyser (Ängelholm, Sweden) apparatus will be used to measure haemoglobin on Day 0 or any other day if clinically warranted.

3.11.3 PCR GENOTYPING PCR genotyping analysis will be performed in order to distinguish true recrudescence (same parasite strain) from a newly acquired infection (different parasite strain). Capillary blood samples for PCR will be collected for all patients at enrolment and during follow-up in case of LCF or LPF after Day 7.

2-3 drops of capillary blood will be collected on FTA cards, stored individually in zip-lock bags with desiccant, and kept away from humidity, excessive heat and light.

The genotyping will be performed at the department of Medical Microbiology, at the Academic Medical Center (Amsterdam, The Netherlands), under the supervision of Prof. Dr Tom van Gool. A material transfer agreement will be signed. The genotyping procedure will be based on comparison of the two-locus genotype resulting from expression of the P. falciparum MSP-1 and MSP-2 gene alleles in pre- (enrolment) and post-treatment (failure) samples27. Pre- and post-treatment pairs with similar genotype will be classified as recrudescence (true failure), and pairs with different genotype will be classified as re-infection.

3.11.4 QUALITY CONTROL OF MALARIA DIAGNOSIS Before the study starts, correct laboratory procedures, such as staining technique, staining time, dilution and data reporting will be established. A blinded re-reading of routine malaria slides (of which at least 20 will be positive) will be performed and discordances reviewed.

An external quality control, with a reference parasitological laboratory, is envisaged at the end of the study on a random sample of 20 positives slides collected between Day 0 and Day 42.

3.11.5 MOLECULAR MARKERS FOR ANTI-MALARIAL DRUG RESISTANCE Currently there are no clear molecular markers associated with decreased susceptibility to ACTs. Therefore we do not anticipate at this moment to study molecular markers of ACT resistance. However a region of chromosome 13 on the P. falciparum genome that is linked to decreased parasite clearance rates in response to ACTs has been identified28. If putative markers of artemisinin resistance are identified in the next 5 years the FTA cards from this study should be made available to the World Wide Antimalarial Resistance Network (WWARN) for analysis. Permission to store the FTA cards at -70⁰C at the Amsterdam Medical Centre, The Netherlands for 5 years after termination of the study, and their use for determination of molecular markers of resistance will therefore be requested in the informed consent forms.

3.12 DATA ANALYSIS 3.12.1 DATA MANAGEMENT All case record forms (CRF) will be double-entered daily using EpiData 3.1 software (Odense, Denmark), merged (with verification of inconsistencies) and analysed using Stata (Stata Corporation, USA) statistical software. An interim analysis of early treatment failure will be carried out once all the participants have reached day 3 and their blood smear results are available. This is to assess at an early stage whether the non-inferiority hypothesis regarding early treatment failure should be rejected. At the end of the study analysis, all CRFs and other source data (consent forms, laboratory registers, screening forms, etc) will be stored securely at the capital level. Data will also be submitted to the WWARN database for the international monitoring of anti-malarial drug resistance. A copy of CRFs will also be stored for at least 5 years at MSF-OCA in Amsterdam. The principal investigator is responsible for keeping all screening forms, the case report form and the completed subject identification code list in a secure location.

3.12.2 ANALYSIS PLAN

* Description of the study : numbers of patients screened, number of patients with a P. falciparum infection, number of patients infected with other Plasmodium species, number of patients excluded (and, if possible, reasons for non-eligibility), numbers of included, randomised and analysable patients
* Validity of the study : results on internal and external laboratory quality control, % of overall non analysable patients and % of overall non analysable patients and % loss to follow-up
* Characteristics of included patients: age, sex, weight-for-height, previous intake of anti-malarials, axillary temperature, parasite density, gametocyte carriage, haemoglobin. Chi-square test will be performed to test the adequacy of randomisation.
* Description of study endpoints: numbers of ETF, LCF, LPF and ACPR at Day 42. Similar outcomes would be assessed at Day 28 for comparison with Day 42 efficacy.
* Adverse events: the proportion of adverse events and serious adverse events in all the patients included in the study for each drug;
* PCR genotyping analysis: number of samples analysed, number of recrudescence episodes and re-infections, number of mixed and undetermined results
* Efficacy estimates: Kaplan-Meier survival analysis methods will be used with and without genotyping adjustment. Patients withdrawn, lost to follow-up or with re-infections are censored from the analysis on that day. Patients with a recurrence of parasitaemia, but with missing or undetermined PCR results should be censored on the last visit when the malaria smear was found to be negative (as it is known that the patient was 'cured' at that point).
* Data analysis: Per-protocol analysis followed by a survival analysis using the Kaplan-Meier method. In addition to the reasons for withdrawal listed above, patients will be considered withdrawn from the analysis if the PCR results are unclassifiable or if the results of PCR indicate that the failure is due to re-infection with P. vivax. P. malariae or P. ovale. The cumulative incidence of success and failure rates at day 28/42, PCR-uncorrected and PCR-corrected for each drug; and the proportion of early treatment failure, late clinical failure, late parasitological failure and adequate clinical and parasitological response at day 28/42, with 95% confidence intervals, PCR-uncorrected and PCR-corrected will be calculated 3.12.3 STUDY REPORT At the end of the study, the principal investigator will submit a report on the study and its main outcome. This report will be shared with the national malaria control programme and the Ministry of Health.

The study results will be presented at appropriate scientific meetings and potentially published in a peer-reviewed journal. Data will also be submitted to the WWARN database for the international monitoring of anti-malarial drug resistance.

Study results will be shared with the community leaders, and in patient meetings. Results will be displayed in lay-language in the health clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 59 months
* Weight ≥ 5 Kg
* Slide-confirmed infection with Plasmodium falciparum only (no mixed infections)
* Asexual parasite density between 2000 and 200000/µl of blood
* Measured axillary temperature ≥ 37.5°C
* Ability to swallow oral medication
* High probability of respecting the follow-up visits (residence within 1 hour walking distance from the OPD, no upcoming travel plans, etc.)
* Informed consent from a parent or caretaker aged at least 18 years.

Exclusion Criteria:

* • General danger signs according to the WHO definition (Appendix 5.1.1)

  * Signs of severe/complicated malaria according to the WHO definition (Appendix 5.1.2)
  * Severe anaemia (haemoglobin < 5 g/dL)
  * Known history of hypersensitivity to any of the study drugs
  * Severe acute malnutrition (as defined by a weight-for-height below -3 Z-score and/or symmetrical oedemas involving at least the feet)
  * Concomitant febrile illness due to causes other than malaria with the potential to confound study outcome (measles, acute lower tract respiratory infection, otitis media, tonsillitis, abscesses, severe diarrhoea with dehydration).
  * Having received already a full course of the treatment (or one of the treatments) under study in the previous 28 days (as indicated by the parent/caretaker). Note that previous incomplete anti-malarial intake of treatments under study, or previous intake of anti-malarials not under study, are not exclusion criteria, but details of any such intake should be recorded carefully.
  * History of hypersensitivity reactions or contra-indications to any medicines being tested.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of children with adequate parasitological clearance after treatment of artesunate-amodiaquine (ASAQ) and artemether-lumefantrine (AL) | 42 days
  In a Kaplan Meyer survival curve it will be shown what the parasitological free period is for children treated with ASAQ or AL, uncorrected for PCR (reinfection and recrudescence) and PCR corrected (recrudescence only).

SECONDARY OUTCOMES:
The proportion of early therapeutic failures, late clinical failures and late parasitological failures in a period of 42 days after treatment initiation | 42 days
Recommendations to MoH on choice of antimalarial first line drugs | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Marit de Wit, MD, MIH, Principal Investigator — Medecins sans Frontieres, Operational Centre Amsterdam

IPD SHARING:
Plan to Share IPD: Yes
Data are available on request in accordance with MSF's data sharing policy: http://fieldresearch.msf.org/msf/handle/10144/306488

REFERENCES:
- [Derived] de Wit M, Funk AL, Moussally K, Nkuba DA, Siddiqui R, Bil K, Piriou E, Bart A, Bahizi Bizoza P, Bousema T. In vivo efficacy of artesunate-amodiaquine and artemether-lumefantrine for the treatment of uncomplicated falciparum malaria: an open-randomized, non-inferiority clinical trial in South Kivu, Democratic Republic of Congo. Malar J. 2016 Sep 6;15(1):455. doi: 10.1186/s12936-016-1444-x. PMID 27599612